CLINICAL TRIAL: NCT05329012
Title: Prospective Case Series to Assess the Handling, Healing and Complications of Using a Titanium Small Fragment Plating System With a New Shape Specifically Adapted to the Distal Ulna
Brief Title: Prospective Case Series to Assess Complications of Using Distal Ulna Locking Plate of I.T.S.
Acronym: DUL-ITS
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: DUL - ITS
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-04

CONDITIONS: Ulna Fractures
MeSH Terms: conditions — Ulna Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DUL treatment group: Patients with unstable ulna fractures will be operated and treated with the Distal Ulna locking plate (I.T.S. company) according to clinical routinal indication.
  Interventions: Device: DUL- Distal Ulna Locking PLate (I.T.S)

INTERVENTIONS:
Device: DUL- Distal Ulna Locking PLate (I.T.S) — The patients are surgical treated with the Distal Ulna locking plate according to standard surgical procedures to treat the unstable distal ulna fractures.

SUMMARY:
Background of the study:

Various studies show that the outcome of unstable distal ulna fractures after open reduction and internal fixation is better than closed reduction. The previous plate system for the distal ulna fractures is applied exclusively on the extensor side. This often leads to irritation of the extensor tendons, as well as problems with pronation and supination. With the new shape of the angle-stable distal ulna plate, the investigator hopes that the stability of the fracture osteosynthesis will remain the same and that it will be better tolerated with regard to the surrounding soft tissue, especially the extensor tendons. In this way, an otherwise practically unavoidable removal of osteosynthesis material could - at least in some cases - be avoided and some patients spared a follow-up operation.

With this in mind, the investigator tries to achieve the greatest possible reconstruction and stability for early functional follow-up treatment with a slightly bulky implant placed in the tendon-free area.

DETAILED DESCRIPTION:
With this study, the application and usability of the new angle-stable plate system should be determined and documented.

New value of the study:

This system enables an optimal position of the plate on the distal ulna, on the one hand due to the position on the flexor side and on the other hand due to the new shape, adapted to the anatomy of the distal ulna. The locking system using angle-stable screws corresponds to the systems previously used by I.T.S.

Design:

Prospectively, handling, advantages and possible complications of the angle-stable, distal ulna plate; Company I.T.S. in the osteosynthesis of the unstable distal ulna fracture. A total of 20 patients with unstable distal ulna fractures are to be treated and evaluated over a period of 12 months according to the study design.

Risk/Benefit:

With the use of the angle-stable distal ulna plate, company I.T.S. the patients broken bone may heal better. However, it is also possible that the patient will not benefit directly from his/her participation in this clinical trial. The Expected Benefit of the Locking Distal Ulnar Plate; Company I.T.S. includes:

* Reduced risk of bone misalignment after surgery.
* Less risk of irritating tendons on the plate with the new location.
* A removal of the osteosynthesis material could possibly be avoided.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. unstable distal ulna fractures

Fracture classification according to Biyani [4]: all types

Exclusion Criteria:

1. Age under 18 years old
2. stable fractures of the ulna
3. Patient had one before ulna fracture
4. Patient may result in physical or intellectual disability consent not grant
5. Patient is for more Check-ups not available (Abroad)
6. Patient does not have full legal capacity
7. Alcohol and drug abuse
8. Increased risk of anesthesia (from ASA 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unstable distal ulna fractures who are over 18 years of age are included in this study. Patients should not have any additional pathology or previous damage to the distal radioulnar joint and should remain available for further examinations (e.g. no tourists, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Complicationsrate | 1 year
  Percentage of complications rate of patients treated with DUL

SECONDARY OUTCOMES:
Clinical outcome (range of motion) | 1year
  Degree of the possible range of motion using a goniometer to measure the movement angles in correlation of the healing process. The better the range of motion the higher the value. Normally the following limits are given:
  Radial: least 0 degree, maximum: 20 degree Ulnar: least 0 degree, maximum: 40 degree Extension: least 0 degree, maximum: 70 degree Flexion: least 0 degree, maximum: 70 degree Pronation: least 0 degree, maximum: 90 degree Supination: least 0 degree, maximum: 90 degree
Clinical outcome (grip strength wrist) | 1year
  Extent of possible grip strength measurement using dynanometer in correlation of the healing process.
  Minimum: 0 kilogram Maximum: 80 kg
Patient Reported Outcome (function) | 1 year
  Percentage of the patients with reduced or normal outcome after fractures using questionnaires like the DASH Score in correlation of the healing process. This is a score reporting the functional outcome, satisfaction and quality of life. Best score is 100%, least score 0%
Patient Reported Outcome (pain) | 1 year
  Percentage of the patients with remaining pain after fracture using the visual analog scale in correlation of the healing process.
  The scale reports about the intensity of pain. The maximum pain and least score is 10, and the best score is 0 which means "no pain".

REFERENCES:
- [Derived] Stock K, Benedikt S, Kastenberger T, Kaiser P, Arora R, Zelger P, Pallua JD, Schmidle G. Outcomes of distal ulna locking plate in management of unstable distal ulna fractures: a prospective case series. Arch Orthop Trauma Surg. 2023 Jun;143(6):3137-3144. doi: 10.1007/s00402-022-04549-4. Epub 2022 Jul 18. PMID 35849186